CLINICAL TRIAL: NCT00273819
Title: Non-Invasive Detection of Revascularizable Cardiomyopathy
Brief Title: Study of Coronary Artery Disease by Two Types of Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AS0006; 00795
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Congestive Heart Failure
Keywords: Congestive heart failure, LV dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

INTERVENTIONS:
Procedure: CT angiography

SUMMARY:
The purpose of this study is to test the ability of a new X-ray technique called CT angiography to identify significant narrowing of the coronary arteries compared to traditional coronary angiogram.

DETAILED DESCRIPTION:
Objective:

In patients with newly diagnosed cardiomyopathy it is the standard of care to perform coronary angiography. This procedure can separate ischemic from non-ischemic cardiomyopathy and identifies patients who may be eligible for revascularization as a therapeutic modality. With the advent of multidectector row-computed tomography technology, it is becoming possible to non-invasively identify significant atherosclerotic stenoses with acceptable sensitivity and specificity. The goal of this study is to compare non-invasive computed tomography (CT) angiography with traditional coronary angiography to identify proximal, and hence revascularizable, coronary artery disease in patients with cardiomyopathy. Revascularizable is defined a 3 vessel proximal disease, left main disease, or left main equivalent disease (ostial left anterior descending and ostial left circumflex).

Research Design:

This study is prospective, interventional, single site with the interpreting radiologists blinded to the results from previous angiography.

Methods:

Subjects will be patients with cardiomyopathy, defined as an ejection fraction less than 40%. Exclusion criteria include known allergy to contrast medium, previous anaphylaxis, and renal insufficiency (serum creatinine greater than 1.5). We would like to enroll 30 patients. After giving informed consent, all eligible patients will undergo CT angiography, performed using new multi-slice technology. The results of previously obtained transthoracic echocardiography and standard coronary angiography will be reviewed. Following CT angiography all patients will have a repeat measurement of serum creatinine to screen for contrast induced nephropathy. Results of the CT angiography will be analyzed to determine sensitivity and specificity for identifying revascularizable coronary artery disease, compared to coronary angiography as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Congestive heart failure with EF<40%
* Age> 18 years

Exclusion Criteria:

* Contrast allergy
* Renal insufficiency
* Inability or unwillingness to sign a consent
* Diabetes Mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2005-10; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Detection of coronary disease by CT angiography

SECONDARY OUTCOMES:
Disease meets latest ACC/AHA guidelines for CABG

CONTACTS AND LOCATIONS:
Overall Officials: Aseem Vashist, M.D., Principal Investigator — VACHS and Yale University School of Medicine; Mehran Sadeghi, M.D., Principal Investigator — VACHS and Yale University School of Medicine
Locations (1):
- VACT Healthcare System-Yale School of Medicine, West Haven, Connecticut, United States